CLINICAL TRIAL: NCT00972465
Title: Phase IIa Study of Nimotuzumab Plus Irinotecan as Second-line Treatment in Metastatic Colorectal Cancer With Wild Type K-ras
Brief Title: Study of Nimotuzumab to Treat Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Shen Lin, Department of GI Oncology,Peking University, School of Oncology, Beijing Cancer Hospital & Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT-CRC-T
Record Dates: First submitted 2009-09-04; First posted 2009-09-07 (Estimated); Last update posted 2009-09-07 (Estimated); Status verified 2009-09

CONDITIONS: Advanced Colorectal Cancer
Keywords: nimotuzumab colorectal cancer chemotherapy
MeSH Terms: interventions — nimotuzumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Nimotuzumab and chemotherapy — Experimental: Nimotuzumab and Irinotecan
  the chemotherapy treatment: Irinotecan (180 mg/m2/time, 1 time/14 days, until disease progression)
  the nimotuzumab treatment: 3 levels (200 mg/w, 400 mg/w, 600 mg/w, weekly, until disease progression)
  Other Names: Nimotuzumab

SUMMARY:
Nimotuzumab is an IgG1 humanized monoclonal antibody that recognized an epitope located in the extra cellular domain of the human epidermal growth factor receptor (EGFR). Clinical efficacy has been shown in adult with head and neck cancer. The study assessed the safety, and efficacy of the combination of Nimotuzumab administered concomitantly with chemotherapy in patients with advanced colorectal cancer.

DETAILED DESCRIPTION:
Nimotuzumab and Irinotecan will be administered to the patient until disease progression or development of toxicity preclude further treatment.Irinotecan will be administered once every 14 days,the dosage is 180mg/m2; Nimotuzumab treatment be divided 3 levels:200mg/w,400mg/w,600mg/w,weekly.The patients'blood test and liver and renal function tests will be monitored weekly, a physical exam and reassessment of the tumor will be performed and every 6 weeks,when the total result is the CR or PR, the result of the 6th and the 12th week should be compared.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed before performing any of the study's specific procedures.
* ECOG performance status 0-2.
* Age > 18，both genders.
* Metastatic colorectal cancer confirmed by pathology, or locally advanced unresectable colorectal cancer, or postoperative recurrence and metastasis colorectal cancer
* Disease progression after receiving oxaliplatin ± fluorouracil in first-line treatment
* At least 1 measurable lesions ,( longest diameter≥ 1 cm by spiral computed tomography (CT) scan or MRI)
* Life expectancy more than 3 months.
* K-ras is wild type
* Use of an effective contraceptive method for patients of both sexes when there is a risk of conception and/or pregnancy.
* Liver metastasis, lesions smaller than 50% of the liver; Lung metastasis, lesions smaller than 30% of the lung
* Haemoglobin≥90g/L , granulocyte≥1.5×109/L ,WBC ≥3×109/L, platelet count≥100×109/L
* TBIL≤ 1.5 x ULN ,ALK≤ 2.5 x ULN or ≤ 5ULN（Liver metastasis），AST and ALT≤ 2.5 x ULN or ≤ 5ULN（Liver metastasis）,Creatinine ≤ 1.5 x ULN
* No brain metastasis

Exclusion Criteria:

* Previous radiotherapy at lesions within three months
* Other first line chemo-agents treatment except oxaliplatin ± fluorouracil
* Received other anti EGFR monoclonal antibody treatment
* Complete or incomplete intestinal obstruction
* Participation in other interventional clinical trials within 1 month
* Psychiatric disease affected cognitive ability, including brain metastasis
* Peripheral neuropathy lesion is more than I stage
* History of serious allergic or allergy
* Pregnant or breast-feeding women
* Patients with the history of Serious lung or hear disease
* Other malignant tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-12 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Safety and toxicity of this new treatment. Both acute and chronic toxicity will be evaluated. | within study period

SECONDARY OUTCOMES:
To determine the complete response rate, partial rate, disease response rate, disease control rate in the patients subject to treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shen Lin, Principal Investigator — Department of GI Oncology,Peking University, School of Oncology, Beijing Cancer Hospital & Institute
Locations (3):
- China (3):
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Peking University, School of Oncology, Beijing Cancer Hospital & Institute, Beijing
  - China People's Liberation Army (PLA)81 Hospital, Nanjing